CLINICAL TRIAL: NCT02132221
Title: Long-term Opioid Therapy in Chronic Pain Patients: Investigation of Tapering Strategies and Impact on Hyperalgesia
Brief Title: Cessation of Long-term Opioid Therapy in Chronic Pain Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment too slow given study timeline
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, James P. Rathmell, MD, Chief, Division of Pain Medicine, Department of Anesthesia, Critical Care and Pain Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Partners IRB 2013P000881
Record Dates: First submitted 2013-10-24; First posted 2014-05-07 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain
Keywords: Chronic non cancer pain; Long term opioid therapy; Side effects; risks; function; negative benefit/risk ratio
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Experimental): cognitive therapy (10 weekly sessions)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- no CBT- wait list (No Intervention): no cognitive therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 10- weekly 1h30 group sessions including psychoeducation and group discussions on pain, pain coping, opioid mechanisms, and relationship between mood, sleep, stress and pain.
  Other Names: CBT; Cognitive therapy; Cognitive therapy workshop
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
This research is being done to better understand how to help patients who are not receiving enough relief from opioid prescription medications for chronic non-cancer pain. Opioids are a group of medications that includes morphine, oxycodone-, hydrocodone-, etc. These medications are also called narcotics. Research has shown that patients not benefiting from their opioid prescription medication often feel better when they stop taking it. However, stopping or reducing pain medications can be a difficult transition. Although they do not have much benefit from their medication, many patients are afraid to stop because they feel these medications are the only things giving them a bit of relief. Different strategies can be used to help patients through the period of tapering and it is not clear which one is best. The investigators will test a specific approach used during regular care in the clinic: cognitive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age above 18.
* Chronic non-cancer pain (pain for 6 or more months, current pain not attributed to a cancerous disease).
* Referrals to the Massachusetts General Hospital (MGH) Center for Pain Medicine for opioid taper.
* Chronic (more than 3 months) prescription of morphine, oxycodone, hydrocodone, hydromorphone, codeine or any formulation of these medications.
* Morphine dose equivalent of 60 mg or above.
* Opioid treatment has to be stable (plus or minus20%) over the last 3 months.
* Meeting Substance Abuse and Mental Health Services Administration (SAMHSA) criteria for exit from chronic opioid therapy
* Willingness to taper and participate in treatment as randomized (including cognitive workshop sessions), able to meet the protocol follow-up schedule and activities
* Agreement to undergo random urine toxicology assays, which will be recommended to prescribing physician during study.
* Agreement to sign an opioid contract, as recommended to prescribing physician.
* Informed consent to study (IRB approved informed Consent form).
* English Language Literacy.

Exclusion Criteria:

* Methadone, suboxone or fentanyl patch: the tapering with these opioids would not be comparable to the other patients. As enrolment will be open during about 12 months, if a patient was motivated to participate in the study, they could be referred to the pain clinic for advice on a switch to a medication that could allow inclusion. They would, 3 months after this switch, become eligible for the study.
* Pregnancy.
* History of epilepsy and drug-induced seizures.
* Proof of current diversion of drugs or recent substance related legal problems (e.g. buying/selling on the streets).
* Concurrent use of illicit drugs and narcotics (urine toxicology), active diagnosis of substance abuse or dependence disorder within last 3 months.
* Absence of the prescribed drug in the urine toxicology
* Refusal of taper or dose reduction trial.
* Preference for suboxone or related treatments.
* Severe psychiatric condition and/or cognitive deficits limiting patient's ability to participate
* Involved in concurrent opioid management for an acute pain condition.
* Current suicidal ideation.
* Severe and unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological or hematological disease.
* General conditions that would impede participation in a group intervention, as assessed by evaluating physician (e.g. cognitive impairment, tendencies towards physical aggression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with daily opioid dose below 50% of initial dose | 10 weeks
  successful taper
signs of hyperalgesia on Quantitative Sensory Testing (QST) | 10 weeks
  evolution of QST scores following taper

SECONDARY OUTCOMES:
signs of hyperalgesia on QST | 24 weeks
  at 3 months follow-up from taper, evolution of hyperalgesia
number of patients who are not prescribed opioids on daily basis ("full taper") | within 10 weeks
  described as not taking opioids on a daily basis
Time to reach >50% taper. | 24 weeks
  time to reach 50% taper will eb recorded in all individuals
Pain scores (Brief Pain Inventory) | 10 and 24 weeks
Absolute opioid dose reduction | 10 and 24 weeks
  calculation of absolute dose reduction
Functional Impairment | 10 and 24 weeks
  Brief Pain Inventory Interference scale and National Institute of Health Patient Reported Outcomes Measurement Information System (PROMIS) scale
Number of patients who reach a full taper amongst those having not reached this outcome at 10 weeks. | 24 weeks
Anxiety and depression (HADS). | 10 and 24 weeks
Withdrawal (COWS measure). | 10 and 24 weeks
Hedonic tone (SHAPS). | 10 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James P Rathmell, MD, Principal Investigator — Department of Anesthesia, Critical Care, Pain Medicine
Locations (1):
- Massachusetts General Hospital Center for Pain Medicine, Boston, Massachusetts, United States